CLINICAL TRIAL: NCT01803152
Title: A Phase I Trial of Dendritic Cell Vaccination for Children and Adults With Sarcoma
Brief Title: Dendritic Cell Vaccine for Children and Adults With Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Macarena De La Fuente, MD (Other)
Responsible Party: Sponsor-Investigator, Macarena De La Fuente, MD, Assistant Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110462
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Sarcoma; Soft Tissue Sarcoma; Bone Sarcoma
Keywords: Metastatic Sarcoma; Relapsed Sarcoma; Dendritic Cell; Myeloid Derived Suppressor Cells; MDSC; MDSC Inhibition
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — lentiviral minigene vaccine of COVID-19 coronavirus; Gemcitabine; Imiquimod; Leukapheresis; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1-DC Vaccine/Lysate (Experimental): * Leukapheresis: Baseline, post-surgery;
  * Dendritic Cells Vaccine (DC Vaccine): Post-Leukapheresis, administered once weekly in dose-escalation scheme for 4 weeks;
  * Lysate of Tumor (Lysate): Post-DC Vaccine therapy, administered during weeks 8, 12, 16 and 20;
  * Imiquimod: Self-applied topically by subject before and after scheduled DC Vaccine or Lysate administrations.
  Interventions: Biological: Dendritic Cells Vaccine; Biological: Lysate of Tumor; Drug: Imiquimod; Procedure: Leukapheresis
- Part 2-Gemcitabine/DC Vaccine/Lysate (Active Comparator): * Leukapheresis: Baseline, post-surgery;
  * Gemcitabine: Post-Leukapheresis, administered once weekly for 3 weeks;
  * Dendritic Cells Vaccine (DC Vaccine): Post-Gemcitabine therapy, Recommended Phase 2 Dose (RP2D) administered once weekly for 4 weeks;
  * Lysate of Tumor (Lysate): Post-DC Vaccine therapy, administered during weeks 12, 16, 20 and 32;
  * Imiquimod: Self-applied topically by subject before and after scheduled DC Vaccine or Lysate administrations.
  Interventions: Biological: Dendritic Cells Vaccine; Biological: Lysate of Tumor; Drug: Gemcitabine; Drug: Imiquimod; Procedure: Leukapheresis

INTERVENTIONS:
Biological: Dendritic Cells Vaccine — Subjects will receive DC Vaccine administered once weekly, via intradermal injection, for 4 weeks for a total of four vaccinations, per study protocol.
  Other Names: DC Vaccine
Biological: Lysate of Tumor — Post-DC Vaccine therapy. Up to 1.5 mg of Lysate of tumor per dose administered via intradermal injection at intervals defined by study protocol.
  Other Names: Lysate; Tumor Lysate
Drug: Gemcitabine — Post-surgery, Leukapheresis and clearance of subject. Gemcitabine 1000 mg/m2 IV will be administered once weekly for 3 weeks per study protocol.
  Other Names: Gemzar
  Arms: Part 2-Gemcitabine/DC Vaccine/Lysate
Drug: Imiquimod — Subjects will self-apply Imiquimod topically to each designated vaccine site before and after scheduled administrations of DC Vaccine or Lysate, per study protocol.
  Other Names: Aldara
Procedure: Leukapheresis — Baseline, post-surgery blood draw via catheter to obtain peripheral blood mononuclear cells (PBMCs) from which Dendritic cells will be obtained.
  Other Names: Pheresis

SUMMARY:
The purpose if this study is to evaluate an investigational vaccine using patient-derived dendritic cells (DC), a type of white blood cell that helps fight infections in the body, (DC) (a vaccine made out of participants' own cells and tumor) to treat sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 1 - 100 years old.
2. Histologically or cytologically confirmed sarcoma either relapsed or without known curative therapies. Both bone sarcomas and soft tissue sarcomas are eligible. Osteosarcoma, chondrosarcoma, Ewing's sarcoma and any other diagnoses of sarcoma are eligible as long as there is soft tissue that can be excised and be used to prepare lysate. Subjects presenting only with lesions that are only comprised of bone are excluded. Any number of prior therapies is allowed, including zero.
3. No radiotherapy to other sites planned and/or other chemotherapy planned for the study period. No radiotherapy or chemotherapy to have been received for at least 4 weeks before first vaccine administration. To allow for better local control without introducing undue toxicity into the trial, brachytherapy at time of surgery scheduled to end by one week before first vaccination is allowed if the radioactive source is to be removed (e.g. catheters can be placed if removable but implanted seeds are not allowed). In the event of positive margins being determined after surgical resection, but not determined in time for the placement of brachytherapy catheters, external beam radiotherapy may start after the last DC vaccination is administered but before the lysate boosts begin, and radiation must be planned to be complete before the first lysate boost.
4. No treatment with corticosteroids, antihistamines or salicylates for at least 1 week before first vaccination.
5. Adequate organ function (to be measured at enrollment)

   * Absolute neutrophil count (ANC) ≥ 0.75* 10^3/µL
   * Lymphocytes ≥ 0.5 * 10^3/µL
   * Platelets ≥ 75 * 10^3/µL
   * Hemoglobin ≥ 9 g/dL
   * Aspartate aminotransferase (AST)/Alanine transaminase (ALT) ≤ 2.5 X upper limit of normal (ULN); if liver metastases, ≤ 5 X ULN
   * Serum Creatinine ≤ 1.5 X ULN
   * Total Bilirubin ≤ 3 X ULN
   * Albumin > 2 g/dL
6. Karnofsky/Lansky score of ≥ 70% or Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Subjects must agree to use adequate method of contraception or abstinence throughout and up to 4 weeks after the study treatment completion.
8. Life expectancy of > 3 months.
9. Written consent by patient or parent(s) (if patient is < 18 years) on an institutional review board (IRB)-approved informed consent form prior to any study-specific evaluation. Assent is required from children as per University of Miami (UM) IRB guidelines. Subject must be capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent.

Exclusion Criteria:

1. Pregnancy
2. Breast feeding females.
3. Any concomitant participation in other therapeutic trials
4. Virus serology known to be positive for HIV (testing is not required in the absence of clinical suspicion)
5. Documented immunodeficiency or autoimmune disease
6. Concomitant treatment with corticosteroids, antihistamines (H1 and H2 inhibitors) or salicylates. Patients may be eligible if the treatment is stopped at least 1 week before the first vaccination.
7. Brain metastases unless they have been stable for 3 months off of treatment directed specifically at them.
8. Known allergy to gemcitabine or its formulation components. Intolerant to gemcitabine

   * Does not apply to cohorts to be treated without gemcitabine
   * Prior therapy with gemcitabine is allowed on all cohorts
9. Refusal to use adequate contraception for fertile patients (females and males) during the study and for 30 days after the last dose of study treatment.
10. Any serious or uncontrolled medical or psychiatric condition that in the opinion of the investigator makes the patient not able to participate in the study.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From Day 1 to 30 Days Post-Treatment, about 9 months
  To demonstrate that DC vaccination loaded with tumor lysate is feasible and that therapy with the vaccine with topical imiquimod (as final step in vaccine maturation), with or without the inhibition of MDSC by gemcitabine pre-treatment, is safe in pediatric and adult subjects with metastatic and refractory sarcoma.

SECONDARY OUTCOMES:
Measurement levels of Myeloid Derived Supressor Cells before and after treatment | From Baseline to 3 Months Post-Treatment, up to 12 months
  To explore biomarkers of immune response. Assessment will include measurement of levels of Myeloid Derived Supressor Cells before and after treatment and T and B cell subsets before and after treatment.
Progression-free survival | Up to 24 months Post-Treatment
  To obtain preliminary clinical benefit by evaluating progression-free survival (PFS)in patients receiving this DC vaccine with or without gemcitabine pre-treatment. PFS is defined as the time elapsed from the start of treatment to the date of documented progression or death, whichever comes first. For surviving patients without progression who begin alternative treatment, PFS will be censored at the last date of documented progression-free status prior to starting alternative treatment. Similarly, losses to follow up will be censored at the last date of documented progression-free status.
Overall Survival | Up to 5 years Post-Treatment
  To obtain preliminary clinical benefit by evaluating overall survival in patients receiving this DC vaccine with or without gemcitabine pre-treatment. Overall survival is defined as the time elapsed from the start of treatment until death. For surviving patients, follow-up will be censored at the date of last contact.
The rate of Complete Response (CR) or Partial Response (PR) in subjects receiving treatment | Up to 24 months Post-Treatment
  To obtain preliminary clinical benefit by evaluating response rate (RR) in patients receiving this DC vaccine with or without gemcitabine pre-treatment. Response will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) Criteria, version 1.1.
Measurement levels of Myeloid Derived Supressor Cells after Gemcitabine treatment | From Baseline to End of Treatment, about 10 months
  To determine if gemcitabine is effective in the inhibition and depletion of Myeloid Derived Supressor Cells in the study patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gina D'Amato, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goff PH, Riolobos L, LaFleur BJ, Spraker MB, Seo YD, Smythe KS, Campbell JS, Pierce RH, Zhang Y, He Q, Kim EY, Schaub SK, Kane GM, Mantilla JG, Chen EY, Ricciotti R, Thompson MJ, Cranmer LD, Wagner MJ, Loggers ET, Jones RL, Murphy E, Blumenschein WM, McClanahan TK, Earls J, Flanagan KC, LaFranzo NA, Kim TS, Pollack SM. Neoadjuvant Therapy Induces a Potent Immune Response to Sarcoma, Dominated by Myeloid and B Cells. Clin Cancer Res. 2022 Apr 14;28(8):1701-1711. doi: 10.1158/1078-0432.CCR-21-4239. PMID 35115306